CLINICAL TRIAL: NCT07218809
Title: A Randomised, Open-label, Phase III Study of AZD5335 Versus Mirvetuximab Soravtansine in FRα-high and AZD5335 Versus Investigator's Choice Chemotherapy in FRα-low Expressing High-grade Platinum-resistant Epithelial Ovarian Cancer Patients (TREVI-OC-01)
Brief Title: AZD5335 vs. Mirvetuximab Soravtansine in FRα-high and AZD5335 vs. Chemotherapy in FRα-low Platinum-resistant Ovarian Cancer
Acronym: TREVI-OC-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: European Network of Gynecological Oncological Trial Groups (ENGOT) (Unknown); GOG Foundation, Inc. (GOG Foundation) (Unknown); Ventana Medical Systems, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D8991C00001
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer; Peritoneal Cancer; Follopian Tube Cancer; Platinum Resistant Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — mirvetuximab soravtansine; Paclitaxel; liposomal doxorubicin; Topotecan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD5335 in FRa-high cohort (Experimental): AZD5335 IV (intravenous) in FRa-high cohort
  Interventions: Drug: AZD5335
- Mirvetuximab Soravtansine (MIRV) in FRa-high cohort (Active Comparator): MIRV AIBW IV in FRa-high cohort
  Interventions: Drug: Mirvetuximab Soravtansine (MIRV)
- AZD5335 in FRa-low cohort (Experimental): AZD5335 IV (intravenous) in FRa-low cohort
  Interventions: Drug: AZD5335
- Investigator´s choice chemotherapy in FRa-low cohort (Active Comparator): Investigator's choice of chemotherapy Paclitaxel IV Pegylated liposomal Doxorubicin (PLD) IV or Topotecan IV in FRa-low cohor
  Interventions: Drug: Paclitaxel; Drug: Pegylated liposomal Doxorubicin (PLD); Drug: Topotecan

INTERVENTIONS:
Drug: AZD5335 — antibody drug conjugate
  Arms: AZD5335 in FRa-high cohort; AZD5335 in FRa-low cohort
Drug: Mirvetuximab Soravtansine (MIRV) — antibody drug conjugate
  Other Names: Elahere
  Arms: Mirvetuximab Soravtansine (MIRV) in FRa-high cohort
Drug: Paclitaxel — chemotherapy
  Other Names: Taxol; Onxol
  Arms: Investigator´s choice chemotherapy in FRa-low cohort
Drug: Pegylated liposomal Doxorubicin (PLD) — chemotherapy
  Other Names: Doxil; Caelyx
  Arms: Investigator´s choice chemotherapy in FRa-low cohort
Drug: Topotecan — chemotherapy
  Other Names: Hycamtin
  Arms: Investigator´s choice chemotherapy in FRa-low cohort

SUMMARY:
The intention of the study is to demonstrate superiority of AZD5335 versus standard of care by assessment of progression-free survival (PFS) in women with high-grade, platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal cancer, expressing high or low FRα levels.

DETAILED DESCRIPTION:
Approximately 1100 adult participants will be enrolled after central FRα testing into two independent cohorts (about 550 FRα-high and 550 FRα-low) and randomized 1:1 within each cohort to receive AZD5335 or the relevant standard of care (mirvetuximab soravtansine in FRα-high; investigator's choice single-agent chemotherapy in FRα-low). Participants will remain on assigned treatment and undergo regular tumor evaluations per RECIST v1.1 until disease progression or another reason for treatment discontinuation.

All participants will be followed for overall survival. An independent data monitoring committee (IDMC) of external experts will periodically review unblinded safety and interim efficacy to confirm participant safety and study integrity.

ELIGIBILITY:
Key Inclusion criteria

* Participants with confirmed diagnosis of high-grade serous EOC, primary peritoneal cancer, or fallopian tube cancer.
* Participants must have platinum-resistant disease:
* Participants who have only had one prior line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response (CR or PR) and then progressed between > 3 months and ≤ 6 months after the date of the last dose of platinum.
* Participants who have received 2 or 3 lines of platinum therapy must have progressed ≤ 6 months after the date of the last dose of platinum.
* Participants must have radiologically progressed on or after their most recent line of therapy.
* Participants must have received at least one, but no more than 3, prior systemic lines of anti-cancer therapy, and for whom single-agent therapy is appropriate as the next line of treatment
* Participants with documented BRCA mutation (germline and/or somatic) must have received prior PARPi if the participant is eligible per approved label and standard-of-care institutional guidelines, except in cases of documented contraindication, precaution or intolerance.
* Provision of an FFPE tumour tissue sample

Key Exclusion criteria

* Participants with endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumours containing any of the above histologies, or low-grade or borderline ovarian tumour.
* Primary platinum-refractory disease, defined as disease that did not respond to or has progressed ≤ 3 months after the last dose of first line platinum-containing chemotherapy.
* Participants with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring
* Current signs, symptoms, or clinical investigations consistent with bowel obstruction, including sub-occlusive disease.
* Participant has non-infectious ILD/pneumonitis or has a history of non-infectious ILD/pneumonitis that required oral or IV steroids or supplemental oxygen, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Prior treatment with any FRα-targeted therapy, including MIRV, or any TOP1i ADC.
* Major surgical procedure within 4 weeks of the first dose of study intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2028-11-17 (Estimated); Study Completion 2030-05-27 (Estimated)

PRIMARY OUTCOMES:
Progression free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from randomization to radiographic progression as assessed by the Investigator per RECIST v1.1, or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.

OTHER OUTCOMES:
Second progression free survival (PFS2) | Up to approximately 5 years
  Time from randomization to second progression or death (PFS2) is defined as the time from randomization to the earliest progression event (following the initial progression) subsequent to the first subsequent therapy, or death.
Objective response date (ORR) | Up to approximately 5 years
  ORR is defined as the proportion of participants who have a complete or partial response, as determined by the investigator, per RECIST v1.1.
Duration of response (DoR) | Up to approximately 5 years
  DoR is defined as the time from the date of first documented response until the date of documented progression per RECIST v1.1, as assessed by the investigator, or death due to any cause.
Health-related Quality of Life (HrQoL) | Up to approximately 5 years
  Change from baseline in selected subscales of EORTC QLQ C30; global health status, physical function and EORTC QLQ OV28 hormonal symptoms (EORTC IL).
CA-125 Response Rate (CA-125 RR) | Up to approximately 5 years
  Proportion of participants achieving CA-125 response per GCIG criteria

CONTACTS AND LOCATIONS:
Locations (104):
- United States (17):
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Evanston, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Towson, Maryland
  - Research Site, Burlington, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, The Bronx, New York
  - Research Site, Dayton, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Fairfax, Virginia
- Australia (8):
  - Research Site, Adelaide
  - Research Site, Auchenflower
  - Research Site, Box Hill
  - Research Site, Campbelltown
  - Research Site, Clayton
  - Research Site, Melbourne
  - Research Site, St Leonards
  - Research Site, Waratah NSW
- Belgium (3):
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Leuven
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Montreal, Quebec
- Chile (3):
  - Research Site, Port Montt
  - Research Site, Santiago
  - Research Site, Viña del Mar
- China (17):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Czechia (3):
  - Research Site, Nový Jičín
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Aarhus, Denmark
- France (7):
  - Research Site, Amiens
  - Research Site, Avignon
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Saint-Herblain
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Tours
- Germany (5):
  - Research Site, Bonn
  - Research Site, Dresden
  - Research Site, Schwäbisch Hall
  - Research Site, Tübingen
  - Research Site, Wiesbaden
- Greece (2):
  - Research Site, Athens
  - Research Site, Pátrai
- India (7):
  - Research Site, Bhubaneswar
  - Research Site, Delhi
  - Research Site, Dhanvantari Nagar
  - Research Site, Kolkata
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, Surat
- Ireland (2):
  - Research Site, Cork
  - Research Site, Dublin
- Israel (6):
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (9):
  - Research Site, Brescia
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
- Japan (3):
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Tsu
- Research Site, A Coruña, Spain
- Research Site, Uppsala, Sweden
- Research Site, Tainan, Taiwan
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
  AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles.
  When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment https://vivli.org/. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/